CLINICAL TRIAL: NCT05733403
Title: Comparison of Hemodynamic Results of Two Different Fluid Managements in Reduction Mammoplasty Operation
Brief Title: Comparison of Hemodynamic Results of Two Different Fluid Managements
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Demet Altun, attending anesthesiologist, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021/588
Record Dates: First submitted 2022-10-28; First posted 2023-02-17 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Perioperative Fluid Management
Keywords: fluid therapy; hemodynamic parameters; The pulse contour cardiac output system; inducible nitric oxide synthetase
MeSH Terms: interventions — Isotonic Solutions; Norepinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stroke Volume Variation (SVV) Group (Active Comparator): When SVV value ≥ 14%, 250cc isotonic will be given within 10min. 250cc isotonic boluses will be repeated until the SVV drops below 14%. If MAP< 65 mmHg despite the SVV falling below 14%, a bolus of 4mcg noradrenaline(NA) will be administered. During the operation, if the SVV is below 14% and the MAP is < 65mmHg, a bolus of 4mcg NA will be administered.
  Intraoperative balance, amount of bleeding, number of fluid boluses and NA administrations, total additional fluid and NA amount, total number of hypotensive episodes will be recorded.
  The times when the breast tissue was removed, the weights of the removed tissues and the amount of bleeding will be recorded.
  Basal and 3 more arterial blood gases will be taken when the breast tissue is removed and early postoperatively, and Hgb, lactate, and base excess values will be recorded. iNOS values in blood will be recorded after basal iNOS and breast tissue are removed.
  The creatinine value will be recorded on the 1st postoperative day.
  Interventions: Drug: isotonic solution; Drug: Noradrenaline
- Mean Arterial Pressure (MAP) Group (Active Comparator): If MAP value under below 65mmHg, 250ml isotonic will be given within 10 min. However, if MAP is still below 65mmHg, a bolus of 4mcg NA will be administered, if no response, 4mcg NA will be repeated. If MAP falls below 65mmHg again, 250 ml isotonic will be administered again in 10 min; if it does not improve, 4mcg of NA will be given iv.
  Intraoperative balance, amount of bleeding, number of fluid boluses and NA administrations, total additional fluid and NA amount, total number of hypotensive episodes will be recorded.
  The times when the breast tissue was removed, the weights of the removed tissues and the amount of bleeding will be recorded.
  Basal and 3 more arterial blood gases will be taken when the breast tissue is removed and early postoperatively, and Hgb, lactate, and base excess values will be recorded. iNOS values in blood will be recorded after basal iNOS and breast tissue are removed.
  The creatinine value will be recorded on the 1st postoperative day.
  Interventions: Drug: isotonic solution; Drug: Noradrenaline

INTERVENTIONS:
Drug: isotonic solution — Isotonic solutions are IV fluids that have a similar concentration of dissolved particles as blood.
  Other Names: 0,9% NaCl
Drug: Noradrenaline — Noradrenaline itself is classified as a sympathomimetic drug: its effects when given by intravenous injection of increasing heart rate and force and constricting blood vessels make it very useful for treating medical emergencies that involve critically low blood pressure.
  Other Names: Norepinephrine

SUMMARY:
In the reduction mammoplasty operations performed in the Plastic and Reconstructive surgery operating room in our clinic, the female patient group, who does not have co-morbidities and does not exceed middle age, is followed by infusion of crystalloid at a constant rate of 4 ml/kg. If the mean arterial pressure (MAP) is <65 mmHg, it is treated with fluid boluses, and in cases where no response is obtained, with noradrenaline boluses. However, in this process, frequent and severe hypotensive episodes are observed, especially after removal of more than a few kilograms of breast tissue. In these hypotensive episodes, factors other than the blood volume lost with the tissue may also play a role. For this reason, we aimed to evaluate the iNOS levels by assuming that the blood levels of "inducible nitric oxide synthetase" (iNOS), which is stored in large amounts in adipose tissues and has been shown to play a role in lipid metabolism, may increase with the manipulation of breast tissue, and accordingly increased nitric oxide may lead to hypotension.

DETAILED DESCRIPTION:
The main purpose of intraoperative fluid therapy is to optimize intravascular volume, mean arterial pressure (MAP) and cardiac output, while ensuring tissue perfusion, while not causing dehydration and fluid overload in the patient. While hypovolemia may cause problems such as organ perfusion disorders and ischemia; Hypervolemia may lead to pulmonary edema, cardiac load, prolonged need for mechanical ventilation and susceptibility to related infections. Although fluid management in the perioperative period has been extensively studied in many studies, a standard practice has not been established. The amount considered restrictive in some studies may be liberal in others. In recent years, the use of dynamic parameters, which are formed as a result of cardiopulmonary interactions and whose high sensitivity and specificity have been proven by many studies, has been increasing day by day for the evaluation of intravascular volume. Pulse pressure variation(PPV) and stroke volume variation(SVV) are two of these dynamic parameters. The pulse contour cardiac output (FloTrac) system, which is a fairly newly developed method that calculates cardiac output and stroke volume directly from the arterial waveform, is used for measurement without the need for calibration.

In the reduction mammoplasty operations performed in the Plastic and Reconstructive surgery operating room in our clinic, the female patient group, who does not have co-morbidities and does not exceed middle age, is followed by infusion of crystalloid at a constant rate of 4 ml/kg. If the mean arterial pressure (MAP) is <65 mmHg, it is treated with fluid boluses, and in cases where no response is obtained, with noradrenaline boluses. However, in this process, frequent and severe hypotensive episodes are observed, especially after removal of more than a few kilograms of breast tissue. In these hypotensive episodes, factors other than the blood volume lost with the tissue may also play a role. For this reason, we aimed to evaluate the iNOS levels by assuming that the blood levels of "inducible nitric oxide synthetase" (iNOS), which is stored in large amounts in adipose tissues and has been shown to play a role in lipid metabolism, may increase with the manipulation of breast tissue, and accordingly increased nitric oxide may lead to hypotension.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteering to participate in the study
2. ASA classification 1 or 2
3. The patients who will undergo reduction mammoplasty operation

Exclusion Criteria:

1. Being under the age of 18 or over the age of 65
2. Presence of serious hypertension

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Cardiac index | during surgery
  Cardiac index (CI) is a haemodynamic parameter that relates the cardiac output (CO) from left ventricle in one minute to body surface area (BSA),thus relating heart performance to the size of the individual. The unit of measurement is litres per minute per square metre (L/min/m2).

SECONDARY OUTCOMES:
Number of bolus administrations of noradrenaline | during surgery
  For the MAP group, if MAP is still below 65 mmHg despite a bolus of 250ml isotonic fluid, a bolus of 4mcg noradrenaline will be administered, if no response, 4mcg noradrenaline will be repeated.
  For the SVV Group, a 4 mcg bolus of noradrenaline will be given if MAP< 65 mmHg despite the SVV falling below 14% with isotonic boluses.
Number of bolus administrations of isotonic fluid | during surgery
  For the MAP group, the number of administrations of 250 ml of isotonic fluid delivered in 10 minutes when MAP < 65 mmHg For the SVV group, the number of administrations of 250 ml of isotonic fluid administered in 10 minutes when SVV≥ 14%
The Number of Hypotensive Episodes | during surgery
  The number of times the MAP value falls below 65mmHg during surgery
Intraoperative Fluid Balance | during surgery
  the difference between the amount of urine output and the amount of bleeding from the amount of fluid given
Plasma iNOS Levels | Up to 6 hours
  difference in serum iNOS levels preoperatively and after removal of mammoplasty material
Lactate value | Up to 6 hours
  Values measured by perioperative arterial blood gas analysis
Base deficit value | Up to 6 hours
  Values measured by perioperative arterial blood gas analysis
Creatinine value | Preoperative and Postoperative 1st day
  Blood level is checked on the preoperative and postoperative 1st day
Urea value | Preoperative and Postoperative 1st day
  Blood level is checked on the preoperative and postoperative 1st day
Hemoglobin value | Preoperative and Postoperative 1st day
  Blood level is checked on the preoperative and postoperative 1st day

CONTACTS AND LOCATIONS:
Overall Officials: Ceren Yılmaz, Resident, Principal Investigator — Istanbul University; Demet Kıvanç, researcher, Principal Investigator — Istanbul University; Ali E Çamcı, Prof., Study Director — Istanbul University
Locations (1):
- Istanbul University, Department of Anesthesiology, Istanbul, Fatih, Turkey (Türkiye)

REFERENCES:
- [Result] Li J, Ji FH, Yang JP. Evaluation of stroke volume variation obtained by the FloTrac/Vigileo system to guide preoperative fluid therapy in patients undergoing brain surgery. J Int Med Res. 2012;40(3):1175-81. doi: 10.1177/147323001204000338. PMID 22906292
- [Result] Anavi S, Tirosh O. iNOS as a metabolic enzyme under stress conditions. Free Radic Biol Med. 2020 Jan;146:16-35. doi: 10.1016/j.freeradbiomed.2019.10.411. Epub 2019 Oct 28. PMID 31672462